CLINICAL TRIAL: NCT06433141
Title: Evaluation of Clinical Performance, Parent's Satisfaction, Gingival Health and Bacterial Effects of Bioflex Crowns & Endocrowns Compared to Ready-Made Zirconia Crowns on Pulpotomized Primary Molars: A Randomized Clinical Trial
Brief Title: Evaluation of Bioflex Crowns Endocrowns Compared to Ready-Made Zirconia Crowns on Pulpotomized Primary Molars
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, kareem ragab abdallah el hosary, head of dental depertment -tanta militery hospital, Al-Azhar University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 966/5604
Record Dates: First submitted 2024-05-12; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Primary Teeth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bio-flex crown (Active Comparator): bio-flex crown will be used as a final restoration for pulp treated primary molar, selection of suitable sized crown , it will be cement with glass ionomer cement after pulpotmy procdure clincal performance, parent satsification ,bacterial adherence will be evaluated with a follow up period 1 year
  Interventions: Procedure: treatment option for primary second molar
- endo-crown (Active Comparator): endo-crown will be used as a final restoration for pulp treated primary molar, after pulpotomy procdure endo-crown preperation design will be done and CAD/CAM, endo crown will be luted according to e-max protocol clincal performance, parent satsification ,bacterial adherence will be evaluated with a follow up period 1 year
  Interventions: Procedure: treatment option for primary second molar
- zirconia crown (Other): zirconia crown will be used as a final restoration for pulp treated primary molar, selection of suitable sized crown after preperation of tooth and use try-in kit to select siutable size ,zirconia is sensitive for blood contamination , it will be cement with glass ionomer cement after pulpotmy procdure clincal performance, parent satsification ,bacterial adherence will be evaluated with a follow up period 1 year
  Interventions: Procedure: treatment option for primary second molar

INTERVENTIONS:
Procedure: treatment option for primary second molar — final restoration for primary second molars

SUMMARY:
This study will be conducted to evaluate clinical performance, parent's satisfaction, gingival health and bacterial effects of Bioflex crowns &Endocrowns compared to ready-made zirconia Crowns on Pulpotomized primary molars

DETAILED DESCRIPTION:
Intervention: Pulptomy Procedures The tooth will be anaesthetized. Then, it will be isolated using a rubber dam. Caries will be removed with a sterile non-end cutting bur # 558 to complete the removal of the pulp chamber roof under copious water coolant spray. Coronal pulp tissue remnants will be removed with a sharp, sterile excavator. A piece of cotton soaked with formocresol will be inserted into the pulp chamber for 5 minutes. After removing the formocresol pellet, a thick mix of zinc- oxide/eugenol paste will be packed into the pulp chamber to seal the oriﬁces.

Restoration of the tooth:

According to the groups restoration will be as the following:

Group A: Endocrowns tooth preparation, scanning, cementation:

For the endocrowns A layer of light -cured glass ionomer cement ° of 1 mm thickness will be applied over the ZOE- to isolate it from the successive resin based restorations and adhesives- leaving a minimum of 3 mm of the pulp chamber to provide an adequate thickness for the endocrown core.

Round-end tapered stone will be used to achieve depth cuts of 1.5 mm for occlusal clearance A wheel stone will complete the occlusal reduction and making butt joint ﬁnish line.

Tapered stone of 8-degree angle will be used to prepare axial wall ﬂared, the pulp chamber walls to a standard degree of divergence.

Abrasive rubber tip will be used to smoothening and rounding the internal angles giving a polished and smoothed preparation.

Endocrown will be manufactured using CAD/CAM technology internal wall of crown will be treated with etchant material, rinsed, dried then silane coupling agent Dual-cure resin cement will be applied on the crown fitting surface for endocrown cementation. Group B: Preformed Bioflex crowns

According to manufacturer instruction the preparation will be as the follow:

Light -cured glass ionomer filling of adequate thickness will be applied over the ZOE to seal the cavity before preparation A digital caliper will be used to measure a mesio-distal dimension of tooth then suitable sized preformed crown will be selected.

Tooth preparation will be carried out with a tapered diamond bur for occlusal reduction by 1-1.5 mm, including the central groove.

The proximal preparation will be around 0.5 mm to clear the contact area Placement of the crown will be achieved by a snug fit followed by contouring using a Hover's plier.

Crown cementation will be carried out using glass ionomer cement and removal of excess cement using floss or explorer.

Group C: performed zirconia crowns Light -cured glass ionomer filling of adequate thickness will be applied over the ZOE to seal the cavity before preparation.

A digital caliper will be used to measure a mesio-distal dimension of tooth then suitable sized preformed crown will be selected.

A diamond bur will reduce the occlusal surface by 1.5-2 mm Interproximal contacts will be prepared with a tapered fissure bur. About 1-2 mm sub gingival preparation will be performed The selected crown will be placed and checked. The passive fit of the crown will be assessed and will be luted with glass ionomer cement.

Consistent firm finger pressure will be applied during cementation. Observations:

Clinical Performance Assessment Retention, marginal adaption, fracture of the restoration were scored using a modified United States Public Health Service (USPHS) criterion.

Dental plaque accumulation and gingival condition were assessed using plaque index (PI) and GI.

Preparation time and cementation assessment using stop watch to record time from preparation start till final restoration cementation.

Clinical performance and oral status will be assessed at follow-up periods of 3 (T1), 6 (T2), and 12 (T3) months. At the end of the follow-up (T3), parent's satisfaction analysis toward the color, shape, and size of three restorations will be adopted to directly evaluate their satisfaction toward their children's restorations. Parents' responses were rated on a 5-point Likert-type scale.Microbiological analysis:

The swabs will be collected before preparation of crowns, 3 months, 6 months and 12 months after cementation. The number of Streptococcus Mutans, lactobacillus will be digitally counted. Swabs will be taken from occlusal surface by means of the tips of sterile cotton The number of Streptococcus Mutans, lactobacillus will be digitally counted. Swabs will be taken from occlusal surface by means of the tips of sterile cotton Samples will be preserved in a transporting medium tube containing 9ml thioglycolate broth medium. All specimens were transported immediately to microbiological lab.

ELIGIBILITY:
Inclusion Criteria:

1 - Parents' and patients' acceptance and cooperation 2- Apparently Healthy children. 3- Child's age ranging from 4 to 8 years old. 4- Primary 2nd molars with deep carious lesion indicated for vital Pulptomy 5- No periapical pathological lesion 6- No root resorption exceeding more than 2/3 of root length.

Exclusion Criteria:

1. Medically compromised children (bleeding disorders, cardiac patient and any systemic diseases could affect oral and gingival health.
2. Presence of para-functional habits. Such bruxism, TMJ disorders
3. Non-restorable tooth.
4. Teeth with non-vital pulp

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
retention of bio-flex crown,zirconia, and endo-crown | follow up will be 3,6,9,12 month
  Retention were scored using a modified United States Public Health Service (USPHS) criterion.
marginal adaptation of bio-flex crown,zirconia, and endo-crown | follow up will be 3,6,9,12 month
  marginal adaptation were scored using a modified United States Public Health Service (USPHS) criterion.
fracture of restoration of bio-flex crown,zirconia, and endo-crown | follow up will be 3,6,9,12 month
  fracture of restoration were scored using a modified United States Public Health Service (USPHS) criterion.
gingival health of bio-flex crown,zirconia, and endo-crown | follow up will be 3,6,9,12 month
  • Dental plaque accumulation and gingival condition were assessed using plaque index (PI) and GI.

SECONDARY OUTCOMES:
parent's satisfaction analysis | follow up will be 3,6,9,12 month
  Parents' responses were rated on a 5-point Likert-type scale.

OTHER OUTCOMES:
Microbiological analysis | follow up will be 3,6,9,12 month
  number of Streptococcus Mutans, lactobacillus will be digitally counted.

CONTACTS AND LOCATIONS:
Overall Officials: kareem elhosary, master degree, Study Chair — Al-Azhar University
Locations (1):
- Faculity of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after 1.5 years

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT06433141/Prot_SAP_000.pdf